CLINICAL TRIAL: NCT03913364
Title: Evaluation of B. Bifidum 900791 as a Modulator of Microbiota, Inflammatory Mediators and Metabolic Hormones in Breast Milk From Obese Mothers
Brief Title: Impact of B. Bifidum 900791 Intake on Breast Milk Characteristics of Obese Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Martin Gotteland, Head, Lab. of Digestive physiology, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UChile-Bifidice-1
Record Dates: First submitted 2019-04-08; First posted 2019-04-12 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Maternal Obesity
Keywords: obesity; breast milk; probiotic; IL-6; CRP; Insulin; Adiponectin; Resistin; breastmilk microbiota; Bifidobacterium
MeSH Terms: conditions — Pregnancy in Obesity; Obesity; Insulin Resistance | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Obese mothers and normal-weight mothers will each be randomized in two groups to receive the probiotic product or the placebo. Colostrum and breastmilk samples will obtained at days 2 and 30 post-partum, respectively, and infant fecal samples at day 30.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Obese mothers (Experimental): One portion (50g) of an ice-cream containing the probiotic B. bifidum 900791 (>10(exp7)/g) every other day during the last month of gestation and the first month of lactation
  Interventions: Dietary Supplement: Probiotic
- Placebo Obese mothers (Placebo Comparator): One portion (50g) of an ice-cream without probiotic every other day during the last month of gestation and the first month of lactation
  Interventions: Dietary Supplement: Placebo
- Experimental normal weight mothers (Experimental): One portion (50g) of an ice-cream containing B. bifidum 900791 (>10(exp7)/g) every other day during the last month of gestation and the first month of lactation
  Interventions: Dietary Supplement: Probiotic
- Placebo normal weight mothers (Placebo Comparator): One portion (50g) of an ice-cream without probiotic every other day during the last month of gestation and the first month of lactation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — B. bifidum 900791-containing ice cream
  Other Names: Bifidice
  Arms: Experimental Obese mothers; Experimental normal weight mothers
Dietary Supplement: Placebo — Placebo ice-cream
  Arms: Placebo Obese mothers; Placebo normal weight mothers

SUMMARY:
Human breast milk harbours a specific microbiota including bacteria from the Lactobacillus and Bifidobacterium genera, that contribute to the bacterial colonization of the infant gut in the post-natal period. An entero-mammary pathway has been suggested by which selected bacteria from the maternal gut would be transmitted to the mammary gland through dendritic cell trafficking by the lymphatic pathway. Accordingly, some studies have detected the presence of probiotic strains in breast milk from mothers who were consuming them. The administration of probiotic supplements to lactating mothers has also been shown to modulate milk concentrations of inflammatory markers and metabolic hormones, impacting positively the infant health. Noteworthily, many of these inflammatory and hormonal biomarkers are altered in the breastmilk from pre-pregnancy obese mothers, compared with these who were normal-weight, possibly affecting the infant health. It is unclear whether the breast milk microbiota of obese mothers is altered and the impact of probiotic administration on the breastmilk microbiota and on the normalization of breastmilk alterations in obese mothers is unknown.

Based on these antecedents, the aim of this study is to determine if the administration of a B. bifidum 900791-containing foodstuff to mothers during the perinatal period normalizes the breast milk concentrations of interleukin (IL)-6, C-Reactive Protein (CRP), insulin, adiponectin and resistin, and the microbiota of obese mothers, compared with normal-weight mothers.

ELIGIBILITY:
Inclusion Criteria:

* Women in their last month of pregnancy, who were normal-weight (18.5<BMI<25kg/m2) or who were obese (BMI>30kg/m2) before pregnancy, and their children

Women recruited should have expressed their wish to have their child through normal delivery, and to breastfeed at least during the first month post-partum.

Exclusion Criteria:

* Women with chronic diseases (type 2 diabetes, renal diseases, autoimmune diseases, tumor, chronic inflammatory diseases, etc.).
* Women with a history of digestive surgery.
* Women whose children are hospitalized more than 24hours in the neonatal unit
* Women who require antibiotic treatment during the perinatal period.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein concentration in breastmilk | Day-30
  Concentration of CRP in breastmilk

SECONDARY OUTCOMES:
IL-6 concentration in breastmilk | Day 30
  Concentration of IL-6 in breastmilk
Insulin concentration in breastmilk | Day 30
  Concentration of Insulin in breastmilk
Resistin concentration in breastmilk | Day 30
  Concentration of resistin in breastmilk
Adiponectin concentration in breastmilk | Day 30
  Concentration of adiponectin in breastmilk
Milk microbiota diversity | Day 30
  Intra-and Interindividual diversity of the milk microbiota
Milk microbiota composition | Day 30
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing
Presence of B. bifidum 900791 in breastmilk | Day 30
  Presence of the probiotic strain B. bifidum 900791 in breastmilk
Infant fecal microbiota diversity | Day 30
  Intra-and Interindividual diversity of the infant fecal microbiota
Infant fecal microbiota composition | Day 30
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing

OTHER OUTCOMES:
Colostrum IL-6 | Day 2
  Concentrations of IL-6 in colostrum
Colostrum CRP | Day 2
  Concentrations of CRP in colostrum
Colostrum insulin | Day 2
  Concentrations of insulin in colostrum
Colostrum resistin | Day 2
  Concentrations of resistin in colostrum
Colostrum adiponectin | Day 2
  Concentrations of adiponectin in colostrum
Colostrum microbiota diversity | Day 2
  Intra-and Interindividual diversity of colostrum
Presence of the probiotic strain in colostrum | Day 2
  Presence of the probiotic strain B. bifidum 900791 in colostrum
Colostrum microbiota composition | Day 2
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing
Presence of mastitis | Days 0-30 pp.
  Presence of mastitis in the mother during the first month post-partum
Presence of infant colic | Days 0-30 pp.
  Appearance of colic in the infant during the first month post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Barrera, PhD, Principal Investigator — Univ. of Chile; Fabien Magne, PhD, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin R, Langa S, Reviriego C, Jiminez E, Marin ML, Xaus J, Fernandez L, Rodriguez JM. Human milk is a source of lactic acid bacteria for the infant gut. J Pediatr. 2003 Dec;143(6):754-8. doi: 10.1016/j.jpeds.2003.09.028. PMID 14657823
- [Result] Qian L, Song H, Cai W. Determination of Bifidobacterium and Lactobacillus in breast milk of healthy women by digital PCR. Benef Microbes. 2016 Sep;7(4):559-69. doi: 10.3920/BM2015.0195. Epub 2016 May 31. PMID 27241905
- [Result] Jimenez E, Fernandez L, Maldonado A, Martin R, Olivares M, Xaus J, Rodriguez JM. Oral administration of Lactobacillus strains isolated from breast milk as an alternative for the treatment of infectious mastitis during lactation. Appl Environ Microbiol. 2008 Aug;74(15):4650-5. doi: 10.1128/AEM.02599-07. Epub 2008 Jun 6. PMID 18539795
- [Result] Abrahamsson TR, Sinkiewicz G, Jakobsson T, Fredrikson M, Bjorksten B. Probiotic lactobacilli in breast milk and infant stool in relation to oral intake during the first year of life. J Pediatr Gastroenterol Nutr. 2009 Sep;49(3):349-54. doi: 10.1097/MPG.0b013e31818f091b. PMID 19525871
- [Result] Dubos C, Vega N, Carvallo C, Navarrete P, Cerda C, Brunser O, Gotteland M. Identification of Lactobacillus spp. in colostrum from Chilean mothers. Arch Latinoam Nutr. 2011 Mar;61(1):66-8. PMID 22097291
- [Result] Cabrera-Rubio R, Collado MC, Laitinen K, Salminen S, Isolauri E, Mira A. The human milk microbiome changes over lactation and is shaped by maternal weight and mode of delivery. Am J Clin Nutr. 2012 Sep;96(3):544-51. doi: 10.3945/ajcn.112.037382. Epub 2012 Jul 25. PMID 22836031
- [Result] Rautava S. Probiotic Intervention Through the Pregnant and Breastfeeding Mother to Reduce Disease Risk in the Child. Breastfeed Med. 2018 Apr;13(S1):S14-S15. doi: 10.1089/bfm.2018.29076.sjr. No abstract available. PMID 29624429
- [Result] Luoto R, Laitinen K, Nermes M, Isolauri E. Impact of maternal probiotic-supplemented dietary counseling during pregnancy on colostrum adiponectin concentration: a prospective, randomized, placebo-controlled study. Early Hum Dev. 2012 Jun;88(6):339-44. doi: 10.1016/j.earlhumdev.2011.09.006. Epub 2011 Sep 25. PMID 21945174
- [Result] Savino F, Fissore MF, Liguori SA, Oggero R. Can hormones contained in mothers' milk account for the beneficial effect of breast-feeding on obesity in children? Clin Endocrinol (Oxf). 2009 Dec;71(6):757-65. doi: 10.1111/j.1365-2265.2009.03585.x. Epub 2009 Mar 19. PMID 19302580
- [Result] Andreas NJ, Hyde MJ, Herbert BR, Jeffries S, Santhakumaran S, Mandalia S, Holmes E, Modi N. Impact of maternal BMI and sampling strategy on the concentration of leptin, insulin, ghrelin and resistin in breast milk across a single feed: a longitudinal cohort study. BMJ Open. 2016 Jul 7;6(7):e010778. doi: 10.1136/bmjopen-2015-010778. PMID 27388351